CLINICAL TRIAL: NCT03279627
Title: Association of Glycemic Control With Comprehension of Discharge Instructions for Diabetes Therapy and Hospital Readmission
Brief Title: Comprehension of Discharge Instructions for Diabetes Therapy and Hospital Readmission
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mary Korytkowski, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO17050222
Record Dates: First submitted 2017-08-18; First posted 2017-09-12 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: inpatient; hypoglycemia; hyperglycemia; hospital readmission; discharge planning
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypoglycemia: This group will be those who experience a BG < 70 mg/dl in the 24-48 hour time period preceding hospital discharge. Study procedures are identical for each group. All participants in this group will be asked to complete the Diabetes Management Questionnaire.
  Interventions: Other: Diabetes Management Questionnaire
- Hyperglycemia: This group will be those who experience a BG > 250 mg/dl in the 24-48 hour time period preceding hospital discharge. Study procedures are identical for each group. All participants in this group will be asked to complete the Diabetes Management Questionnaire.
  Interventions: Other: Diabetes Management Questionnaire
- Glycemic control: This group will be those who maintain BG of 70 to 250 mg /dl in the 24-48 hour time period preceding hospital discharge. Study procedures are identical for each group, but study outcomes including comprehension of discharge instructions and 1 and 3 month readmissions will be analyzed according to group category.All participants in this group will be asked to complete the Diabetes Management Questionnaire.
  Interventions: Other: Diabetes Management Questionnaire

INTERVENTIONS:
Other: Diabetes Management Questionnaire — Patients will be asked questions regarding their understanding of instructions for home diabetes management within 48 hours of hospital discharge. At 1 and 3 months, participants will be contacted to obtain information regarding ER visits or hospital readmissions.

SUMMARY:
The purpose of this study is to identify and explore the existing components of discharge planning provided to patients with insulin treated diabetes in the inpatient setting and to examine the contribution of glycemic excursions as well as comprehension of discharge instructions among patients with diabetes, in predicting hospital readmissions.

DETAILED DESCRIPTION:
Background: Diabetes is a major contributor to hospital readmissions and health care expenditures. Previous studies have attempted to identify risk factors for readmission among patients with diabetes. However, no studies have looked at some potentially important factors including duration of diabetes, HbA1c, glycemic excursions preceding hospital discharge, and patient comprehension of discharge instructions provided for home diabetes management. In this study, we propose to examine patient understanding of instructions for insulin therapy provided at the time of hospital discharge as a potential risk factor for readmission during the following 30- and 90-day time periods. In addition, we will examine the contribution of glycemic excursions obtained in the 48-hour period prior to discharge on patient understanding of insulin therapy and risk for readmission.

Purpose: The purpose of this study is to identify and explore the existing components of discharge planning provided to patients with insulin treated diabetes in the inpatient setting and to examine the contribution of glycemic excursions as well as comprehension of discharge instructions among patients with diabetes, in predicting hospital readmissions.

Methods: This will be a prospective non-blinded observational study enrolling non-critically ill, non-pregnant, hospitalized patients aged 18-90 years of age with insulin treated diabetes and no evidence of baseline cognitive. The participants will be recruited from August 2017 to December 2018 from the Inpatient Endocrine and Diabetes Consult Services and from daily reports of patients experiencing BG< 70 mg/dL and >300 mg/dL. Eligible participants will be called within 24-48 hours following hospital discharge at which time they will be asked to complete a Diabetes Management Questionnaire to determine their comprehension of the recommendations provided for home-insulin and other diabetes therapies. This questionnaire will include questions about the types of insulin being used, the doses administered, and times given. Patient interviews will be conducted again via a telephone follow up at approximately 30- and 90-days following discharge with specific questions on home blood glucose control and ER or hospital visits and/or readmissions. The Clinical and Translational Science Institute at the University of Pittsburgh will be consulted for statistical analysis.

Study significance:

This study has the potential to identify modifiable factors that can potentially contribute to the observed frequency of hospital readmissions among patients with insulin treated diabetes. This study could also advocate for discharge protocols and close follow up of patients with insulin-treated diabetes following discharge to ensure appropriate understanding of discharge instructions for insulin therapy and home diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-critically ill, hospitalized patients aged 18-90 years with insulin treated diabetes in the hospital

Exclusion Criteria:

* Patients admitted with primary diagnosis of hypoglycemia, DKA; or Hyperglycemic Hyperosmolar Syndrome; patients receiving intravenous narcotic medications; patients discharged to skilled nursing facilities; patients with cognitive impairment defined as dementia or delirium documented in the Electronic Medical Record (EMR); patients with limited life expectancy as determined by "Do Not Resuscitate" Status, or documentation of receiving palliative care or terminal diagnoses with expected survival of less than 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill adult patients with diabetes will be recruited during a period of hospitalization for non-critical illness.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Patient understanding of discharge instructions for home diabetes therapy according to presence or absence of hypoglycemia (defined as BG < 70 mg/dl), hyperglycemia (defined as BG > 250 mg/dl), or BG 70-250 mg/dl at time of hospital discharge | within 48 hours of hospital discharge
  Participants will be asked to complete a questionnaire regarding their home diabetes medications including timing, adjusting, and medication names.

SECONDARY OUTCOMES:
Association between patient understanding of home diabetes therapy and frequency of ER visits and hospital readmissions at 30- and 90-day following the index hospitalization | 1 and 3 months following index hospitalization
  Questionnaire for ER visits and Hospital Readmission

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Korytkowski, MD, Principal Investigator — Univesity of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data with other researchers

REFERENCES:
- [Derived] Patel N, Swami J, Pinkhasova D, Karslioglu French E, Hlasnik D, Delisi K, Donihi A, Siminerio L, Rubin DJ, Wang L, Korytkowski MT. Sex differences in glycemic measures, complications, discharge disposition, and postdischarge emergency room visits and readmission among non-critically ill, hospitalized patients with diabetes. BMJ Open Diabetes Res Care. 2022 Mar;10(2):e002722. doi: 10.1136/bmjdrc-2021-002722. PMID 35246452